CLINICAL TRIAL: NCT01983943
Title: Effects of Hydroxytyrosol on Vascular Health
Brief Title: Olive Oil and Cardiovascular Health
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Invasive Cardiologist, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 13-001080
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Cardiovascular Disease; Endothelial Function
MeSH Terms: conditions — Cardiovascular Diseases | interventions — 3,4-dihydroxyphenylethanol; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroxytyrosol (Experimental): Hydroxytyrosol, the major polyphenol in olive oil, 40mg will be taken once per day for 6 months.
  Interventions: Dietary Supplement: Hydroxytyrosol, the active ingredient in olive oil.; Behavioral: Nutrition counseling; Device: Endopat
- Placebo (Placebo Comparator): Placebo 40mg will be taken once per day for 6 months.
  Interventions: Dietary Supplement: Placebo; Behavioral: Nutrition counseling; Device: Endopat

INTERVENTIONS:
Dietary Supplement: Hydroxytyrosol, the active ingredient in olive oil. — A 40mg capsule will be taken once daily for 6 months.
  Arms: Hydroxytyrosol
Dietary Supplement: Placebo — A 40mg placebo will be taken once per day for 6 months.
  Arms: Placebo
Behavioral: Nutrition counseling — Nutrition counseling on eating a healthy diet will be offered once at baseline.
Device: Endopat — An endopat test will be administered twice, once and baseline and once after 6 months of supplementation, to test endothelial function. This is a non-invasive test that takes about 15 minutes.

SUMMARY:
The purpose of this study is to conduct a double-blind, randomized controlled trial (RCT), to determine if six month supplementation of olive oil can improve the health of the blood vessels and improve long term health of the heart and blood vessels, in patients requiring percutaneous coronary intervention (PCI).

ELIGIBILITY:
Subjects will be included if they have all of the following

1. Age ≥ 18 years old
2. Have known diagnosis of coronary artery disease
3. Demonstrated endothelial dysfunction (reactive hyperemia - EndoPAT score < 2.0) at time of screening

Patient exclusion criteria:

Patients will be excluded if they have one or more of the following:

1. Hypertension (at Screening): any patient with systolic blood pressure (SBP) ≥ 170 mmHg or diastolic blood pressure ≥ 110 mmHg, or hypotension (SBP < 100 mmHg)
2. Uncontrolled Diabetes Mellitus
3. Experienced an acute coronary syndrome within 3 months
4. PCI or revascularization for an acute coronary syndrome within 3 months
5. Second (II) or third (III) degree heart block without a pacemaker and/or concurrent potentially life threatening arrhythmia or other uncontrolled arrhythmia
6. Congestive heart failure NYHA class III and IV
7. Unstable serum creatinine (>2.0)
8. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the olive oil including, but not limited to, any of the following:

   * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
   * Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
   * Evidence of hepatic disease as determined by a history of hepatic encephalopathy, a history of cirrhosis, esophageal varices, or a history of portocaval shunt
9. Any concurrent life threatening condition with a life expectancy less than 2 years
10. History or evidence of drug or alcohol abuse within the last 12 months
11. History of hypersensitivity to any of the study drugs or to medications belonging to the same therapeutic class as the study drugs as well as known or suspected contraindications to the study drugs
12. History of noncompliance to medical regimens or unwillingness to comply with the study protocol
13. History of malignancy other than basal cell skin cancer within the past five years
14. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
15. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
16. Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety
17. Persons directly involved in the execution of this protocol
18. Pregnant or nursing (lactating) women
19. Women of child-bearing potential unless postmenopausal for at least one year, surgically sterile or using effective methods of contraception as defined by local Health Authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 6 months
  In order to address these hypotheses, our specific aims are to investigate the effect of administration of six months of hydroxytyrosol in individuals with multiple cardiovascular risk factors and with known coronary artery disease, on: Improvement of endothelial function as determined by peripheral endothelial function testing and circulating EPCs.
Surrogate markers | 6 months
  In order to address these hypotheses, our specific aims are to investigate the effect of administration of six months of hydroxytyrosol in individuals with multiple cardiovascular risk factors and with known coronary artery disease, on: Improvement and normalization of surrogate markers of CVD such as leukocytes, glucose, lipids, renal function, and high-sensitivity C-reactive protein (hs-CRP).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States